CLINICAL TRIAL: NCT02599272
Title: Effects of Mixed Spices on Cardiometabolic Function - the PolySPice (PSP) Study
Acronym: PSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2015/00729
Record Dates: First submitted 2015-10-23; First posted 2015-11-06 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Cardiometabolic Risk
MeSH Terms: interventions — Vegetables

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rice with vegetables but no added spice (Other): Control session - rice with control vegetables (tomatoes and aubergines) - no mixed spices
  Interventions: Other: Rice with tomatoes and peeled aubergine (no spice)
- Rice with vegetables and low spice (Active Comparator): Dose 1 mixed spice session - rice with 6 g powdered mixed spices and 40 g polyphenol rich vegetables (onions, ginger and garlic)
  Interventions: Other: Rice with vegetables and low spice
- Rice with vegetables and high spice (Active Comparator): Dose 2 mixed spice session - rice with 12 g powdered mixed spices and 80 g polyphenol rich vegetables (onions, ginger and garlic)
  Interventions: Other: Rice with vegetables and high spice

INTERVENTIONS:
Other: Rice with tomatoes and peeled aubergine (no spice) — Dose 0
  Arms: Rice with vegetables but no added spice
Other: Rice with vegetables and low spice — Dose 1, Rice with mixed spices (turmeric, coriander, cumin, gooseberry cayenne pepper, cinnamon, clove), tomatoes, peeled aubergine, onion, ginger and garlic
  Arms: Rice with vegetables and low spice
Other: Rice with vegetables and high spice — Dose 2, Rice with mixed spices (turmeric, coriander, cumin, gooseberry cayenne pepper, cinnamon, clove), tomatoes, onion, ginger and garlic
  Arms: Rice with vegetables and high spice

SUMMARY:
The study will investigate whether having mixed spices rich in polyphenols can improve postprandial cardiometabolic response in healthy Chinese men.

DETAILED DESCRIPTION:
Spices have been used for centuries to enhance food flavouring and to maintain health. Use of spices as a culinary ingredient is common amongst people of all ethnicities within South and East Asia. Spices are also one of the main sources of polyphenols in the Asian diet. Several in vitro studies and some in vivo studies, mainly in animals have shown that individual spices, including turmeric (containing curcumin), cinnamon (cinnimic acid), ginger, garlic etc. have been shown to improve glucose and lipid metabolism.However, well-controlled randomised trials, within the normal dietary context in humans are limited.

This study will be conducted using a three-way randomised crossover design using the Latin square approach. In the two treatment sessions, each volunteer will consume a mixed spice dish at two doses (i.e., 'small portion' or 'large portion' curry sauce), and rice as the base ingredient. In the control session, the same base ingredient (rice) but without the mixed spices will be served. The total amount of mixed spices consumed, to be made from dried powders of turmeric, cumin, coriander, gooseberry (amla), cinnamon, clove and cayenne pepper, will be 6 g and 12 g for small and large portion curries respectively. In addition, as added vegetables, the curry meals will contain tomato, garlic, onion and ginger, whereas the control meal will just have tomato and peeled aubergine, although, the total amount of vegetables will remain the same across all dishes (treatment or control).

The primary objective of this study will be to measure postprandial and fasting changes in blood glucose, insulin, triglycerides (TG), free fatty acids (FFA), 24h ambulatory blood pressure (BP), endothelial function and inflammatory markers following consumption of increasing doses of mixed spices in a single meal, on separate occasions.

The secondary objective of the study will be to monitor changes in blood levels of gut hormones, plasma and urine metabolome including polyphenols such as benzoate and hippurate, gut microflora content and function, as a result of the mixed spice intake. A subset of the treatments (control and high spice dose only) will also have interstitial glucose monitored continuously for a period of up to 3 days using the continuous glucose monitoring system (CGMS).

ELIGIBILITY:
Inclusion Criteria:

* Chinese Male
* Age between 21 to 40 years
* Body Mass Index between 18.5 to 27.5 kg/m2
* Waist circumference ≤ 90cm
* Fasting blood glucose < 6.0mmol/L
* Blood pressure <140mmHg systolic or < 90mmHg diastolic
* Do not partake in sports at the competitive and/or endurance levels and willing to stop any strenuous activity during or within 72 hours of test days

Exclusion Criteria:

* Smoking
* Allergic/intolerant to any of the test foods mentioned above, or any of the following common food and ingredients: eggs, fish, milk, peanuts, and tree nuts, shellfish, soya, wheat, gluten, cereal, fruits, dairy products, meat, vegetable, sugar and sweetener, natural food colourings or flavourings, etc.
* Have difficulty passing motion
* Have or had diarrhea in the past 1 month of study participation
* Have any metabolic or cardiovascular diseases (e.g., diabetes, heart condition) or any other diseases involving the small intestine or the colon (e.g., irritable bowel syndrome, inflammatory bowel disease, gastric reflux) Have any liver or kidney disorders or any family history of kidney stones
* Taking any prescribed medication or dietary supplements which may interfere with the study measurements, including consumption of probiotic drinks or supplements, taking antibiotics, laxatives or antidiarrheal medicines likely to interfere with study findings
* Excessive alcohol consumption: consuming alcohol on > 4 days per week with ≥ 6 alcoholic drinks per week
* Individuals who have donated blood within the previous 6 months

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Postprandial changes in interstitial glucose concentration | Up to 48 hours from baseline, taken every 5 minutes
  Postprandial changes in interstitial glucose concentration using continuous glucose monitoring (CGM) following consumption of increasing doses of mixed spices in a single meal
Postprandial changes in plasma insulin concentration | Up to 48 hours from baseline
  Postprandial changes in plasma insulin concentration following consumption of increasing doses of mixed spices in a single meal
Postprandial changes in plasma triglyceride concentration | Up to 48 hours from baseline
  Postprandial changes in plasma triglyceride concentration following consumption of increasing doses of mixed spices in a single meal
Postprandial changes in plasma free fatty acid (FFA) concentration | Up to 48 hours from baseline
  Postprandial changes in plasma free fatty acid (FFA) concentration following consumption of increasing doses of mixed spices in a single meal
Postprandial changes in plasma interleukin-6 (IL-6) concentration | Up to 48 hours from baseline
  Postprandial changes in plasma IL-6 concentration following consumption of increasing doses of mixed spices in a single meal
Postprandial changes in plasma inter-cellular adhesion molecule (ICAM-1) concentration | Up to 48 hours from baseline
  Postprandial changes in plasma inter-cellular adhesion molecule (ICAM-1) concentration following consumption of increasing doses of mixed spices in a single meal

SECONDARY OUTCOMES:
Monitor changes in blood levels of glucagon like peptide 1 (GLP-1) | Up to 48 hours from baseline
  Monitor changes in blood levels of glucagon like peptide 1 (GLP-1) as a result of the mixed spice intake
Monitor changes in blood levels of glucose dependent insulinotropic peptide (GIP) | Up to 48 hours from baseline
  Monitor changes in blood levels of GIP as a result of the mixed spice intake
Monitor changes in blood levels of peptide YY (PYY) | Up to 48 hours from baseline
  Monitor changes in blood levels of PYY as a result of the mixed spice intake
Monitor changes in plasma metabolome (metabolomics) | Up to 48 hours from baseline
  Monitor changes in plasma metabolome including benzoate and hippurate as a result of the mixed spice intake
Monitor changes in urine metabolome (metabolomics) | Up to 48 hours from baseline
  Monitor changes in urine metabolome including hippurate and benzoate as a result of the mixed spice intake
Monitor changes in gut microbiome | Up to 2 days before and up to 8 days after baseline
  Stool samples will be collected at baseline (3 days and 1 day before) and up to 7 days following consumption of curry (1, 3 and 7 days after collection)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

REFERENCES:
- [Derived] Haldar S, Pakkiri LS, Lim J, Chia SC, Ponnalagu S, Drum CL, Henry CJ. Reductions in Postprandial Plasma Allantoin Concentrations With Increasing Doses of Polyphenol Rich Curry Intake - A Randomized Crossover Trial. Front Physiol. 2019 Jan 9;9:1899. doi: 10.3389/fphys.2018.01899. eCollection 2018. PMID 30687117